CLINICAL TRIAL: NCT00827047
Title: A Prospective Randomized Controlled Trial of Total Hemihepatic Vascular Exclusion in Hepatectomy in Hepatocellular Carcinoma Treatment
Brief Title: Total Hemihepatic Vascular Exclusion in Hepatectomy in Hepatocellular Carcinoma Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-012
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Surgical resection; total hemihepatic vascular exclusion; occlusion; bleeding; overall survival
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bites and Stings; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Total Hemihepatic Vascular Exclusion (Active Comparator): Patients with HCC received Total Hemihepatic Vascular Exclusion in hepatectomy.
  Interventions: Procedure: Total hemihepatic vascular exclusion
- Hemihepatic vascular Clamping (Experimental): Patients with HCC received Hemihepatic vascular Clamping in hepatectomy.
  Interventions: Procedure: Hemihepatic vascular Clamping
- Pringle's Maneuver (Experimental): Patients with HCC received Pringle's Maneuver in hepatectomy.
  Interventions: Procedure: Pringle's Maneuver

INTERVENTIONS:
Procedure: Total hemihepatic vascular exclusion — A long vascular clamp is inserted along the midline of the anterior surface of the vena cava,proceed cranially up to the space between the right and the middle hepatic vein trunks. Two tapes are seized with the clamp passing between the anterior surface of the IVC and the liver parenchyma.One tape is use to pass around the hepatic parenchyma for occlusion of the bleeding from the remnant liver;the other is used to loop the right (or left )hepatic vein trunk and short hepatic vein,as well as inferior right hepatic vein,if present. Selectively interrupts the arterial and portal inflow to the part of the liver (right or left hemiliver)ipsilateral to the lesion that requires resection.Thus total hemihepatic vascular exclusion is achieved.
  Other Names: THHVE group
  Arms: Total Hemihepatic Vascular Exclusion
Procedure: Hemihepatic vascular Clamping — Selectively interrupts the arterial and portal inflow to the part of the liver (right or left hemiliver)ipsilateral to the lesion that requires resection. Selective clamping can be achieved after carefully dissecting the right from the left hilar branches or after inserting a clamp between the right and left hilar branches without prior hilar dissection and looping the right or left portal structures with a tape.
  Other Names: Hemihepatic vascular Clamping group
  Arms: Hemihepatic vascular Clamping
Procedure: Pringle's Maneuver — Hepatic pedicle clamping is performed by encircling the hepatoduodenal ligament with a tape and then applying a tourniquet or a vascular clamp until the pulse in the hepatic artery disappears distally.
  Other Names: Pringle's Maneuver group
  Arms: Pringle's Maneuver

SUMMARY:
Total hemihepatic vascular exclusion(THHVE),completely isolates the right or left hemiliver ipsilateral to the lesion that requires resection from the systemic circulation,has the advantage of preventing backflow hemorrhage or air embolism without having to resort to caval blood flow interruption of THVE.This study is to evaluate if THHVE can raduce bleeding,reduce the incidence of complications and improve the patient's free survival and overall survival compared with hemihepatic vascular clamping and Pringle maneuver.

DETAILED DESCRIPTION:
The amount of blood loss and blood transfusion in Hepatectomy have a detrimental effect on the prognosis for Hepatocellular carcinoma(HCC).Intraoperative bleeding remains a major concern during liver resection. The most often used hepatic vascular control methods at present are hepatic pedicle occlusion(Pringle maneuver), hemihepatic vascular clamping,segmental vascular clamping and total hepatic vascular exclusion (THVE).However,all these methods have shortcomings. Pringle maneuver cannot prevent bleeding from hepatic veins and leads to ischemia-reperfusion injury of the liver; Hemihepatic vascular clamping cannot prevent bleeding from hepatic veins as well, and from the remnant (nonoccluded) liver. THVE is a technically demanding technique that requires surgical and anesthetic expertise and may lead to hemodynamic intolerance as well as increased morbidity and hospital stay. Total hemihepatic vascular exclusion(THHVE),completely isolates the right or left hemiliver ipsilateral to the lesion that requires resection from the systemic circulation,has the advantage of preventing backflow hemorrhage or air embolism without having to resort to caval blood flow interruption of THVE.

The purpose of this study is to evaluate if THHVE can raduce bleeding,reduce the incidence of complications and improve the patient's free survival and overall survival compared with other occlusion methods.

ELIGIBILITY:
5Inclusion Criteria:

* Understanding and being willing to sigh the informed consent form.
* Aged 18-75years.
* Corresponding to diagnostic standards of HCC, without any adjuvant therapy,tumor or multiple tumors located in right or left liver lobe.
* The function of heart, lung ,renal is well,without any surgery contraindication.
* KPS score≥60分
* Liver function in the Child-Pugh classification is A or B.
* Tumor AJCC stage isⅠorⅡ.

Exclusion Criteria:

* cannot be follow-up
* liver function in the Child-Pugh classification is C.
* with tumor thrombus in the hepatic vein or main trunk of portal vein
* with extrahepatic metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overall survival and disease free survival | 1,2,or 3 years

SECONDARY OUTCOMES:
Bleeding and blood transfusion ,hepatic function of patients after surgery, the incidence rate of complications | 1,2,or 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, M.D, Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China